CLINICAL TRIAL: NCT07225608
Title: The Acute Effects of Liquid IV's Multi-Ingredient Pre-Workout Supplement, on Endurance, Strength, Energy, and Cognition: A Randomized Crossover Study
Brief Title: The Acute Effects of Liquid IV's Pre-Workout Supplement on Muscle Endurance & Strength, Energy, and Cognition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00089370
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Physical Performance; Exercise Performance; Endurance Exercise; Perceived Exertion; Mood; Energy
Keywords: physical performance; exercise performance; endurance exercise; perceived exertion; strength endurance; mood; energy; L-theanine; Rhodiola Rosea; Creatine

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, crossover study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprietary pre-workout supplement (Experimental): Liquid IV pre-workout supplement powder
  Interventions: Dietary Supplement: proprietary pre-workout supplement
- Control treatment (Placebo Comparator): inactive/inert placebo mixture
  Interventions: Dietary Supplement: Control placebo

INTERVENTIONS:
Dietary Supplement: proprietary pre-workout supplement — proprietary pre-workout supplement
  Arms: proprietary pre-workout supplement
Dietary Supplement: Control placebo — inactive/inert placebo mix
  Arms: Control treatment

SUMMARY:
The goal of this study is to learn if a new pre-workout supplement can improve exercise performance in healthy adults. It will also look at how the supplement affects mood and energy levels.

The main questions it aims to answer are:

Does the pre-workout supplement improve endurance and strength during exercise?

Does it reduce how hard exercise feels (perceived exertion)?

How does it affect participants' mood and energy?

Researchers will compare the pre-workout supplement to a placebo (a look-alike powder that contains no active ingredients) to see if it works.

Participants will:

Take the pre-workout supplement or a placebo before exercise in two separate sessions;

Complete exercise tests after taking each one;

Report how they feel during and after exercise, including mood, energy, and effort.

By bridging gaps in existing research, this study aims to establish a robust scientific foundation for the application of this novel pre-workout supplement in enhancing exercise outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-55
* Must be recreationally trained or trained/developmental as previously defined (McKay et al., 2021)
* Able to read and write in English
* Willing to maintain their regular supplement routine during the study (other than what is listed in exclusion criteria)
* Are not consistently taking, or will discontinue consuming other pre-workout supplements or dietary supplements, such as creatine, rhodiola, L-Theanine, glycerol, stimulants other than caffeine, or ingredients which may promote hydration or enhance physical performance within the past 2-weeks, and throughout the duration of the study.
* Willing to restrict caffeine for 24 hours prior to testing
* Will not participate in any strenuous exercise for a minimum of 72 hours prior to exercise performance assessments. Strenuous exercise as defined for this study includes ½ and full marathons (or more), heavy (i.e.,>80% 1RM) lifting, and any high intensity, physical activity that could make your muscles sore.

Exclusion Criteria:

* Sedentary: Individuals performing less than 150 minutes of moderate or 75 minutes of vigorous activity per week and engaging in resistance training fewer than 2 days per week, with no structured exercise routine.
* Highly trained/national level or professional athlete: Individuals training ≥5 days per week in structured programs, including NCAA Division II/III athletes, national/professional competitors, or those targeting top 20% sport-specific performance norms.
* Known diagnosis of any cardiovascular, metabolic, endocrine, or renal disease
* Recent musculoskeletal injury (<3-months)
* Recent orthopaedic surgery (<12-months)
* History or current malignancy
* Previous gastrointestinal surgery within the past 12 months
* Regular smoker
* Regular drinker (>14 drinks per week)
* Current respiratory infection (i.e. cold) or high temperature (fever) within the past 4-weeks
* Presently using GLP-1 medications
* Individuals with cardiovascular, metabolic, or musculoskeletal disorders;
* Those regularly using anti-inflammatory drugs within the last 4-weeks
* Current use of prescription medications that may influence adaptation to exercise (hormone therapies, peptides, etc.)
* Current consistent chronic use (within the past 2 weeks) of creatine, rhodiola, L-Theanine, glycerol, or other products which contain any of these ingredients.
* Current consistent chronic use (within the past 2 weeks) of stimulants other than caffeine
* Current consistent chronic use (within the past 2 weeks) of ingredients that may promote hydration or enhance physical performance.
* Allergies to study-related materials
* Any condition that may impair their ability to complete the required exercises (determined during screening).
* Female subjects must not be pregnant or lactating
* Are unable to provide informed consent or are non-English speakers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Aerobic Endurance (Graded Cycling Test VO₂max ) | From baseline 70 minutes after treatment consumption, then again on day 6, 70 minutes post treatment consumption
  Participants will complete a graded cycling test on a calibrated cycle ergometer to assess aerobic performance. Maximal oxygen consumption (VO₂max) will be noted if a plateau is observed. using a metabolic cart to determine VO₂max.VO₂max represents the highest rate of oxygen consumption achieved during the test. Proper cycle ergometer setup, including seat height and handlebar position, will be standardized for all participants. Testing will be conducted by trained technicians for consistency.
Local Muscular Endurance (Bench Press to Failure) | From baseline 50 minutes post treatment consumption, then again on day 6, 50 minutes post treatment consumption
  Participants will complete bench press assessments to evaluate muscular strength and endurance. A 5-repetition maximum (5RM) protocol will be used to determine maximal bench press strength. For muscular endurance, participants will complete two sets of bench press at 60% of their 1RM, performing repetitions to fatigue with 2 minutes of rest between sets. Total work volume will be calculated as the product of sets × repetitions. Proper spotting and form supervision will be ensured throughout.
Aerobic Endurance (Graded Cycling Test VO₂peak) | From baseline 70 minutes after treatment consumption, then again on day 6, 70 minutes post treatment consumption
  Participants will complete a graded cycling test on a calibrated cycle ergometer to assess aerobic performance. Oxygen consumption (VO₂) will be continuously monitored every 15 seconds using a metabolic cart to determine VO₂peak. Peak oxygen consumption will be recorded as the highest oxygen uptake value observed during the incremental test. Proper cycle ergometer setup, including seat height and handlebar position, will be standardized for all participants. Testing will be conducted by trained technicians for consistency.
Aerobic Endurance (Graded Cycling Test Time to Exhaustion) | From baseline 70 minutes after treatment consumption, then again on day 6, 70 minutes post treatment consumption
  Participants will complete a graded cycling test on a calibrated cycle ergometer to assess aerobic performance. The total duration in minutes participants are able to sustain the incremental cycling workload until volitional fatigue is recorded. This measures endurance capacity during the graded test. Proper cycle ergometer setup, including seat height and handlebar position, will be standardized for all participants. Testing will be conducted by trained technicians for consistency.
Aerobic Endurance (Graded Cycling Test Total Work Performed) | From baseline 70 minutes after treatment consumption, then again on day 6, 70 minutes post treatment consumption
  Participants will complete a graded cycling test on a calibrated cycle ergometer to assess aerobic performance. Total work (kJ) will be calculated as Σ(power × time)/1000, where power = kp × 50 RPM × 6.118.. This reflects overall exercise performance. Proper cycle ergometer setup, including seat height and handlebar position, will be standardized for all participants. Testing will be conducted by trained technicians for consistency.

SECONDARY OUTCOMES:
Thayer Activation-Deactivation Adjective Checklist (ADACL) | From baseline, 10 minutes pre treatment consumption, then 35 minutes after treatment consumption, and then again 90 minutes post treatment consumption. Until repeated on day 6.
  The Thayer ADACL is a 20-item self-report scale used to assess participants' current mood states across four subscales: Energetic Arousal, Tense Arousal, Calmness, and Fatigue. Participants indicate the extent to which each adjective describes their current state on a 4-point scale ranging from 1 ("definitely feel") to 4 ("definitely do not feel"). Higher scores on Energetic Arousal and Calmness indicate greater energy and calmness, while higher scores on Tense Arousal and Fatigue indicate greater tension and fatigue. Two items, "wide-awake" and "wakeful," are reverse-scored as part of the Fatigue subscale to ensure that higher subscale scores consistently reflect greater fatigue. Subscale scores are analyzed individually to evaluate changes in mood and energy/fatigue responses to supplementation.
Samn-Perelli Visual Analog Scale (VAS) | From baseline, 10 minutes pre treatment consumption, then 35 minutes after treatment consumption, and then again 90 minutes post treatment consumption. Until repeated on day 6.
  The Samn-Perelli VAS is a single-item scale used to assess participants' subjective levels of alertness and fatigue. Participants mark a point along a 7-point scale, where 1 indicates "fully alert" and 7 indicates "completely exhausted." Higher scores reflect greater fatigue or lower alertness. This measure allows quantification of perceived fatigue before and after supplementation, and changes from baseline are used to evaluate the intervention's effects.
Caffeine Visual Analog Scale (VAS) | From baseline, 10 minutes pre treatment consumption, then 35 minutes after treatment consumption, and then again 90 minutes post treatment consumption. Until repeated on day 6.
  The Caffeine VAS is a multi-item visual analog scale used to assess participants' perceived alertness, fatigue, and potential side effects related to caffeine intake. Participants indicate their current state by marking a point along a 100-mm horizontal line, where 0 represents "not at all" and 100 represents "extremely." Scores are recorded in millimeters from the left anchor, with higher values indicating greater intensity of the measured state. Each item is scored separately, and changes from baseline are used to evaluate the effects of supplementation.
Muscle Strength and Strength Endurance (Isometric Mid Thigh Pull) | From baseline 40 minutes after treatment consumption, then again on day 6, 40 minutes post treatment consumption
  Maximal lower-body strength will be assessed using a calibrated isometric mid-thigh pull device. Participants will perform a single maximal effort pull while maintaining standardized body posture and hand placement on the bar. Peak force output, measured in Newtons, will be recorded as the primary indicator of lower-body strength. All tests will be administered by the same technician to ensure procedural consistency.
Lower Body Power and Force Generation (Maximal Countermovement Jump) | From baseline 45 minutes after treatment consumption, then again on day 6, 45 minutes post treatment consumption
  The force plate platform consists of two force plates (left & right) containing four force sensors which measure ground reaction force. The sensors are connected to a laptop and analyzed using Mechanography GRFP Research Edition® software (version 4.2-b05.53-RES). Subjects will perform three maximal vertical CMJs on a calibrated force plate. Subjects will be instructed to stand upright on the center of the force plate with feet shoulder-width apart and hands placed on the hips. Subjects will perform a maximal effort vertical jump with proper form and instructed to land with soft knees and remain still after each jump for data capture. A 30sec rest period will be provided between each trial. Data will be used to assess maximum force output (Fmax), rate of force development (RFD), jump height (inches), and maximum power (Pmax). Force curves will be reviewed for each trial, and results averaged. This will quantify full-body mechanical power under standardized, reproducible conditions.
Body Hydration Bioelectrical Impedance Analysis (InBody) | From baseline, 20 minutes pre treatment consumption, then 30 minutes after treatment consumption, and then again 100 minutes post treatment consumption. Until repeated on day 6.
  Hydration and body water distribution will be assessed using bioelectrical impedance analysis. Parameters include total body water (TBW), extracellular water (ECW), and intracellular water (ICW). Participants will be instructed to arrive in a fasted state, and measurements will be taken under standardized conditions to determine body hydration levels. These values provide insight into overall hydration and fluid compartment balance.
Muscle Strength and Endurance (Grip Strength) | From baseline 35 minutes post treatment consumption, then again on day 6, 35 minutes post treatment consumption
  Handgrip strength will be evaluated using a calibrated hand grip dynamometer. Participants will perform three maximal isometric contractions with their dominant hand, with 30 seconds of rest between attempts. The highest recorded value (in kilograms of force) will be used for analysis. This assessment provides an index of upper-body muscular strength.
Body Hydration (Urine Specific Gravity) | From baseline, 20 minutes pre treatment consumption, then again 100 minutes post treatment consumption. Until repeated on day 6.
  Urine specific gravity will be measured using a handheld refractometer to assess acute hydration status. Participants will provide a midstream urine sample, and the specific gravity value will be recorded to the nearest 0.001. Lower values indicate greater hydration, while higher values suggest increased concentration or dehydration.
  Time Frame: Assessed at baseline and post-supplementation testing.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sikorski, PhD, Principal Investigator — Applied Science and Performance Institute
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No